CLINICAL TRIAL: NCT05305261
Title: Maternal to Neonatal Transmission Antibody Covid-19 Study - The TRAB CoV-19
Brief Title: Mother to Child Transmission of Antibody to Covid-19 The TRAB CoV-19 Study.
Status: Completed | Type: Observational
Sponsor: National University of Malaysia (Other)
Collaborators: Malaysia Automotive Robotics and Innovation of Technology Institute (Unknown)
Responsible Party: Principal Investigator, Rahana Abd Rahman, Associate Professor, National University of Malaysia
Other Study IDs: FF-2021-362
Record Dates: First submitted 2022-03-29; First posted 2022-03-31 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Antibody; Vaccine; Maternal; Cord
Keywords: Covid-19; antibody; pregnancy
MeSH Terms: conditions — Cone-Rod Dystrophies; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Biospecimen Retention: Samples Without DNA — Maternal and cord blood samples taken to measure the antibody levels for Covid-19 at delivery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective clinical study aiming to investigate on the transplacental antibody transmission post Covid-19 infection during pregnancy.

DETAILED DESCRIPTION:
Covid -19 infection has been a significant public health burden as it shifted the paradigm of infectious diseases aiming to control the spread and enhance public immune protection. The introduction of Covid -19 vaccination in December 2020 aimed to combat the infection, thus tremendously helping to flatten the disease worldwide. Channeling the vaccine for the obstetrics field is one of the hallmark strategies to reduce maternal morbidity and mortality. The efficacy of vaccination for the pregnant lady has been established. However, fetus protection via transmission of the antibody during pregnancy is still uncertain. Therefore, this study aims to consolidate further evidence of transplacental antibody post-maternal vaccination aiming for fetal protection following delivery.

ELIGIBILITY:
Inclusion Criteria:

* term pregnancies at 37 weeks or more
* vaccinated 2 doses
* in labour

Exclusion Criteria:

* unvaccinated
* preterm labour less than 37 weeks
* multiple pregnancies

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All vaccinated pregnant women at term with or without a history of covid-19 infection admitted in labour
Sampling Method: Non-Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2021-07-29 (Actual); Primary Completion 2022-03-18 (Actual); Study Completion 2022-03-18 (Actual)

PRIMARY OUTCOMES:
Maternal to Neonatal Transmission Antibody Covid-19 Study - The TRAB CoV-19 | 30 minutes after delivery
  Quantification of Covid-19 antibody levels in maternal and cord blood samples

CONTACTS AND LOCATIONS:
Locations (1):
- UKM Medical Center, Kuala Lumpur, W.Persekutuan, Malaysia

IPD SHARING:
Plan to Share IPD: No